CLINICAL TRIAL: NCT02157532
Title: Intra-arterial Thrombectomy as an Acute Treatment Intervention for Stoke: the Endovascular Acute Stoke Intervention (EASI) Trial
Brief Title: Endovascular Acute Stroke Intervention Trial - the EASI Trial
Acronym: EASI
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Sites are not recruiting.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE 12.224
Record Dates: First submitted 2014-06-02; First posted 2014-06-06 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stroke, Acute
Keywords: Severe stroke; IV tPA; mechanical thrombectomy
MeSH Terms: conditions — Stroke | interventions — Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Best standard treatment (Active Comparator): intravenous r-tPA or any other medical management
  Interventions: Drug: Best standard treatment
- Mechanical thrombectomy (Active Comparator): Endovascular mechanical thrombectomy with stent-retrievers
  Interventions: Procedure: mechanical thrombectomy

INTERVENTIONS:
Procedure: mechanical thrombectomy — Mechanical thrombectomy using any already approved stent-retriever device
  Arms: Mechanical thrombectomy
Drug: Best standard treatment — Intravenous r-tPA infusion or any other medical management option
  Other Names: Medical management
  Arms: Best standard treatment

SUMMARY:
Stroke constitutes the primary cause of acquired disability in adults and the second cause of dementia following Alzheimer disease. It has been shown that patients with a moderate to severe clinical score have occlusion of brain large vessels, resulting in a worse clinical outcome. Many studies have demonstrated that early recanalization after IV rtPA is more restricted, the larger and more proximal the artery. Several systems for mechanical intracranial arterial thrombectomy of large trunks have recently been proposed and are now available. Potential advantages of these mechanical systems on chemical thrombolysis are speed (a few minutes versus 1 hour) and absence of thrombolytic injection.

The objective of the EASI trial is thus to:

* To validate intra-arterial thrombectomy use during the acute phase of cerebral stroke in patients treated with IV thrombolysis or in patients for whom thrombolysis is contra-indicated.
* To determine whether a combined approach, standard treatment plus thrombectomy, is superior to standard treatment alone within 5 h of the appearance of symptoms, in patients with occlusion of proximal cerebral arteries following moderate to severe stroke (NIHSS larger than or equal to 8), evaluated at 3 months.

The design is a randomized, controlled multicentric trial, with a parallel comparison between standard and combined (standard plus thrombectomy) treatment.

480 patients fulfilling eligibility criteria will be sufficient to demonstrate the primary hypothesis of a 15% difference in number of subjects with a favorable mRS (less than or equal to 2) at 3 months, with the assumption of a 25% efficacy for IV thrombolytic treatment at 3 months.

IV thrombolysis is carried out according to standard practice. Mechanical thrombectomy is carried out with already approved devices, according to the manufacturer's instructions, following a diagnostic cerebral angiography.

The primary efficacy endpoint is clinical: favorable mRS (less than or equal to 2) at 3 months.

The primary safety endpoint is rate of death at 3 months and rate of symptomatic hemorrhage at 24 hours.

If the primary hypothesis is validated, expected benefits of this study is a higher rate of autonomy for stroke patients with all the attendant consequences: reduction in hospital stays, and a faster return to the activities of daily life.

DETAILED DESCRIPTION:
Background Stroke constitutes the primary cause of acquired disability in adults and the second cause of dementia following Alzheimer disease. The burden of disease may be substantial since 25% of the victims of stroke are younger than 65 years. Standard treatment is IV rtPA thrombolysis, within 3-4.5 hours of first signs. It has been shown that patients with a moderate to severe clinical score (NIHSS more than 10) have occlusion of proximal large vessels, resulting in a more adverse clinical outcome. Many studies have demonstrated that early recanalization after IV rtPA is more restricted, the larger and more proximal the artery. Recanalization of large arteries occurs more frequently and earlier (leading to better prognosis) with arterial than with venous access. Biochemical arterial treatment appears thus of greater efficacy in terms of recanalization of large vessels, but more inconvenient with respect to setup delays. Several systems for mechanical intracranial arterial thrombectomy of large trunks have recently been proposed and are now available. Results of short case series and prospective multicentric non randomized studies appear favorable. The thrombus obstructing the artery is reached by endovascular means and mechanically removed with the result that orthograde blood flow is re-established in the cerebral territory involved in the ischemia. Potential advantages of these mechanical systems on chemical thrombolysis are speed (a few minutes versus 1 hour) and absence of thrombolytic injection. Mechanical thrombolysis should thus lead to better results than injection of an arterial thrombolytic agent, as well as increase the time window for treatment. In addition, hemorrhagic complications should be reduced.

Objectives

In situations where IV rtPA thrombolysis is not optimal, that is in presumed embolic occlusions of large intracranial arterial trunks (terminal carotid, initial segment of the MCA, distal third of the basilar trunk) with a moderate to severe clinical state (NIHSS greater or equal to 8) and in situations when IV rtPA may be contra-indicated:

* To validate intra-arterial thrombectomy use during the acute phase of cerebral stroke in patients treated with IV thrombolysis or in patients for whom thrombolysis is contra-indicated.
* To determine whether a combined approach, standard treatment plus thrombectomy, is superior to standard treatment alone within 5 h of the appearance of symptoms, in patients with occlusion of proximal cerebral arteries following moderate to severe stroke (greater or equal to 8), evaluated at 3 months.

Design EASI is a randomized, controlled multicentric trial, with a parallel comparison between standard and combined (standard plus thrombectomy) treatment. All adults presenting less than 5 hours after the beginning of symptoms with an NIHSS greater or equal to 8 discordant with imaging data are eligible. Occlusion site, when available, includes intracranial carotid artery, M1 segment of middle cerebral and basilar artery.

480 patients fulfilling eligibility criteria will be sufficient to demonstrate the primary hypothesis of a 15% difference in number of subjects with a favorable mRS (greater than 2) at 3 months, with the assumption of a 25% efficacy (mRS less or equal to 2) for IV thrombolytic treatment at 3 months.

Randomization may take place any time following admission, including during IV thrombolysis. The choice of early randomization, without knowledge of the clinical or angiographic results of IV thrombolysis fulfils several objectives: allow timely delivery of a proven treatment; prevent unnecessary exposure to angiography risks; set up thrombectomy as fast as possible for a maximal efficacy.

IV thrombolysis is carried out according to standard practice. Mechanical thrombectomy is carried out with already approved devices, according to the manufacturer's instructions, following a diagnostic cerebral angiography.

Follow-up includes brain imaging and the mRS at 3 months.

Endpoint measures include:

* Clinical endpoints as measured by the neurologist, and include the NIHSS at baseline and the mRS at 3 months.
* Safety data: complications, death at 3 months, hemorrhage according to 24 hours CT scan.

The primary efficacy endpoint is clinical: favorable mRS (less than or equal to 2) at 3 months.

The primary safety endpoint is rate of death at 3 months and rate of symptomatic hemorrhage at 24 hours.

Secondary efficacy endpoints include:

* Comparison of ASPECTS score between baseline and 24 hours CT scans
* In thrombectomy group, blood flow in treated territory as measured by a TICI reperfusion score of 2 or 3 at end of treatment.

Secondary safety endpoints include

* Rate of hemorrhage on 24 hours CT scan
* Frequency and severity of complications of standard treatment
* Frequency and severity of arterial complications in thrombectomy group
* Frequency and severity of complications at puncture site in thrombectomy group

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* NIHSS greater than or equal to 8
* onset of symptoms is less than 5 hours OR symptom/imaging mismatch
* suspected occlusion of the M1 or M2 segment of the MCA, supraclinoid ICA, or basilar trunk.

Exclusion Criteria:

* established infarction of the target symptomatic territory
* co-morbid diseases which suggest a poor 90 day outcome irrespective of management
* radiologic evidence of hemorrhagic transformation of the infarcted territory

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2013-01; Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
clinical (efficacy): favorable modified Rankin Score (less than or equal to 2) | 3 months
  The efficacy of mechanical thrombectomy compared to standard stroke treatment will be evaluated using the modified Rankin scale score at 3 months. This measure includes the rate of death within 3 months
Rate of symptomatic intracranial hemorrhage | 24 hours
  the incidence of symptomatic hemorrhage on non-contrast CT at 24 hours will be recorded

SECONDARY OUTCOMES:
Infarct evolution | 24 hours
  the evolution of the infarct on CT will be carried out according to a semi-quantitative evaluation using the ASPECT score between the pre-treatment CT and the 24 hour cross-sectional imaging study
Angiographic outcome in patients allocated to mechanical thrombectomy | 2 hours
  In patients allocated to the mechanical thrombectomy arm, the occlusion state of the target vessel will be assessed at the end of the intervention according to the TICI scale
Frequency and Severity of complications | 3 months
  All Adverse Events
Rate of intracranial hemorrhage | 24 hours
  The incidence of hemorrhage on non-contrast CT at 24 hours will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jean Raymond, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM); Serge Bracard, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - Centre Hospitalier de l'Université de Montréal - Hôpital Notre Dame, Montreal, Quebec

REFERENCES:
- [Derived] Poppe AY, Jacquin G, Stapf C, Daneault N, Deschaintre Y, Gioia LC, Odier C, Labrie M, Nehme A, Nico L, Roy D, Weill A, Raymond J. A randomized pilot study of patients with tandem carotid lesions undergoing thrombectomy. J Neuroradiol. 2020 Nov;47(6):416-420. doi: 10.1016/j.neurad.2019.08.003. Epub 2019 Sep 26. PMID 31563589
- [Derived] Khoury NN, Darsaut TE, Ghostine J, Deschaintre Y, Daneault N, Durocher A, Lanthier S, Poppe AY, Odier C, Lebrun LH, Guilbert F, Gentric JC, Batista A, Weill A, Roy D, Bracard S, Raymond J; EASI trial collaborators. Endovascular thrombectomy and medical therapy versus medical therapy alone in acute stroke: A randomized care trial. J Neuroradiol. 2017 Jun;44(3):198-202. doi: 10.1016/j.neurad.2017.01.126. Epub 2017 Feb 24. PMID 28238522